CLINICAL TRIAL: NCT06312904
Title: Effects of Paravertebral Block on Postoperative Analgesia in Children Undergoing Lateral Incision Cardiac Surgery With Cardiopulmonary Bypass: a Randomized Controlled Trial
Brief Title: Paravertebral Block for Postoperative Analgesia in Children Undergoing Lateral Incision Cardiac Surgery With CBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jingfei Guo, Attending Physician, Department of Anesthesiology, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-GSP-QN-7
Record Dates: First submitted 2024-02-29; First posted 2024-03-15 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain
Keywords: Postoperative analgesia; paravertebral block; pediatric cardiac surgery; enhanced recovery after surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paravertebral block group (Experimental): This group of patients will undergo postoperative paravertebral block.
  Interventions: Procedure: paravertebral block
- local infiltration group (Active Comparator): This group of patients will undergo postoperative local infiltration anesthesia.
  Interventions: Procedure: Local infiltration anesthesia

INTERVENTIONS:
Procedure: paravertebral block — After cardiac surgery, the anesthesiologist will use 3mg/kg of 0.375% ropivacaine to conduct paravertebral block.
  Arms: paravertebral block group
Procedure: Local infiltration anesthesia — After cardiac surgery, the anesthesiologist will use 3mg/kg of 0.375% ropivacaine to conduct local infiltration anesthesia.
  Arms: local infiltration group

SUMMARY:
This study aims to compare the effect of paravertebral block and local infiltration anesthesia on postoperative analgesia in children undergoing lateral incision cardiac surgery with cardiopulmonary bypass. The researchers hope to investigate whether children who undergo paravertebral block experience less postoperative pain, have fewer postoperative complications, and recover more quickly.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6-14 years old;
2. Children who have atrial septal defect or ventricular septal defect scheduled for lateral incision cardiac surgery with cardiopulmonary bypass;
3. Inform consent signed by the parent or legal guardian.

Exclusion Criteria:

1. Patients who were intubated, on mechanical circulatory support, or with intravenous inotropes before surgery;
2. Emergency surgery or redo cardiac surgery;
3. Body weight more than 50kg;
4. Diagnosed as severe pulmonary hypertension;
5. Left ventricular ejection fraction less than 45% in most recent echocardiography before surgery;
6. Allergic to ropivacaine or other regular anesthetics, analgesics or other medications regularly used in the study;
7. Preoperative platelet counts less than 100*109/L, coagulopathy or bleeding tendency ;
8. Preoperatively using antiplatelets or anticoagulants;
9. Diagnosed with scoliosis or other contraindications for PVB.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
opioid consumption during the first 24h after surgery | 24 hours postoperatively
  the total amount of sufentanil and other opioids will be calculated as morphine equivalent dose (MED) divided by body weight

SECONDARY OUTCOMES:
FPS-R scale recorded at 6, 12, 18 and 24h postoperatively | 24 hours postoperatively
  The Faces Pain Scale-Revised (FPS-R) is a self-report measure of pain intensity developed for children. It was adapted from the Faces Pain Scale to make it possible to score the sensation of pain on the widely accepted 0-to-10 metric. The scale shows a close linear relationship with visual analog pain scales across the age range of 4-16 years. The bedside nurse will show the patients a picture of six faces, and score 0, 2, 4, 6, 8, and 10 from left to right. "0" equals "no pain" and "10" equals "very much pain." They will ask the patient to choose a face that represents their current pain condition and record the pain score.
The rate of opioid treatment for remedial analgesia between groups | 24 hours postoperatively

OTHER OUTCOMES:
Length of postoperative mechanical ventilation | through study completion, an average of 2 weeks
Length of ICU/hospital stay | through study completion, an average of 2 weeks
The incidence of respiratory depression | through study completion, an average of 2 weeks
  The respiratory depression is defined as: with no obvious upper respiratory tract obstruction: SpO2 < 90% and lasts for more than one minute, or respiratory rate < 8 times/min, or SpO2 < 94% and respiratory rate < 10 times/min, or supplemental oxygen is needed to maintain SpO2 > 94%.
The rate of postoperative nausea and vomiting (PONV) during the 24h postoperatively | through study completion, an average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jingfei Guo, Study Chair — Fuwai Hospital, National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The original data will be published in 2025 on http://www.medresman.org.cn
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2025.1-2026.1
URL: http://www.medresman.org.cn

REFERENCES:
- [Derived] Guo J, Tian L, Kang W, Jia Y, Yuan S. Effects of paravertebral block on postoperative analgesia in children undergoing unilateral thoracotomy cardiac surgery with cardiopulmonary bypass: protocol for a randomised controlled trial. BMJ Open. 2024 Nov 7;14(11):e086462. doi: 10.1136/bmjopen-2024-086462. PMID 39510785

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT06312904/Prot_SAP_ICF_000.pdf